CLINICAL TRIAL: NCT05900414
Title: Pilot Clinical Trial of the Risk Assessment and Personal Preference to Improve Decisions in Atrial Fibrillation Patient Decision Aid for Stroke Prevention in Atrial Fibrillation: the RAPID AFib Pilot Trial.
Brief Title: RAPID AFib Decision Aid for Stroke Prevention in Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Stephen B. Wilton, Associate Professor, Cardiac Sciences, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB22-1737
Record Dates: First submitted 2023-06-04; First posted 2023-06-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: patient decision aid; stroke; shared decision aid; anticoagulant therapy
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (Experimental): Receives web-based information and access to patient decision aid before clinic visit
  Interventions: Behavioral: Electronic patient decision aid
- Control (Active Comparator): Receives web-based information only before clinic visit
  Interventions: Other: Information

INTERVENTIONS:
Behavioral: Electronic patient decision aid — Link to website with information about atrial fibrillation treatments, plus access to the web-based patient decision aid to enable shared decision making between patients and their physicians for atrial fibrillation stroke prevention treatments
  Arms: Patient Decision Aid
Other: Information — Link to website with information about atrial fibrillation treatments
  Arms: Control

SUMMARY:
The goal of this pilot clinical trial is to evaluate the utility of a new electronic patient decision aid for stroke prevention therapy in patients with atrial fibrillation. The main questions it aims to answer are:

Is the patient decision aid acceptable to both patients and physicians? Does the patient decision aid lead to more effective shared decision-making than standard care among patients with atrial fibrillation who are considering stroke prevention therapy? Participants with a recent diagnosis of atrial fibrillation will be enrolled before an upcoming specialist physician visit. Researchers will compare a pre-visit intervention consisting of standard educational materials plus use of the patient decision aid to educational materials alone to see if using the decision aid results in improved shared decision making during the clinic visit.

DETAILED DESCRIPTION:
Background:

Atrial fibrillation (AF) leads to a 4-fold increased risk of stroke, accounting for 15-20% of the 50,000 strokes suffered by Canadians each year. The annual stroke risk in untreated patients is 4.5%, but varies 10-fold based on risk factors captured in clinical prediction tools. Given that oral anticoagulation (OAC) reduces stroke risk by 65%, the majority of AF-associated strokes are potentially preventable. All current Canadian and international AF guidelines strongly recommend use of clinical prediction rules to assess stroke risk, and anticoagulation of high-risk patients. However, population-based studies continue to document significant rates of risk-discordant stroke prevention therapy. Addressing this care gap is a major knowledge translation challenge.

Patient decision aids are knowledge translation tools that can facilitate a process of shared decision-making to improve patient knowledge and decision quality. These tools have the potential to improve both initial therapy selection and adherence, ultimately reducing the risks of AF-associated stroke and unnecessary bleeding. We have developed and performed initial user testing for a new, web-based decision aid, called Risk Assessment and Personal preferences to Improve Decisions for Atrial Fibrillation (RAPID AFib). The tool has 3 sequential functions: (1) it estimates an individual's risk for stroke and for bleeding using published risk scores; (2) it allows them to interactively compare OACs to select one or more therapies that best matches their risk profile and individual preferences ; and (3) it summarizes the risk information and their selected therapy to facilitate discussion with their physician in a Summary Report. This study represents the next step in this program of research, by performing a formal evaluation of the performance of this tool in a real-world clinical setting.

Primary Objective:

To conduct a pilot study to establish the acceptability of the RAPID AFib tool and its impact on the process of shared decision-making for stroke prevention therapy in patients with recent onset AF

Hypothesis:

The RAPID Afib decision aid will be acceptable for both patients and clinicians, and will lead to more effective shared decision-making than standard care among patients with AF who are considering OAC.

Methods:

Study Design: Prospective, randomized pilot study.

Study procedures:

Clinic staff will screen referred patients, then the research team will approach them to confirm eligibility, request informed consent for participation, and collect baseline demographic and clinical data. Consenting patients will be randomized 1:1 using a web-based application linked to the study database to receive the study intervention or control. Randomization will be stratified by clinic site.

All patients will be invited to review an evidence-based website providing information about AF and its management.

Intervention group: Patients randomized to the RAPID AFib intervention will be sent a link to the decision aid website and asked to complete the decision aid before their upcoming visit. They will also be asked to bring the Summary Report to their upcoming clinic visit. A copy of the Summary Report will be added to the patient chart for clinician review.

Control group: Patients randomized to the control group will attend their clinic visit as scheduled, with no further direction from the study team.

Follow-up: Study participation will end after completion of a post-visit survey.

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular AF diagnosed within 12 months, with any level of stroke risk assessed by CHA2DS2-VASc score.
* Age 18 or older
* Either no OAC treatment or treated for less than 90 days.
* Initial specialist AF visit scheduled in 7-30 days.

Exclusion Criteria:

* Valvular AF, defined, per Canadian Cardiovascular Society Guidelines, as AF in the presence of mechanical heart valves, rheumatic mitral stenosis, or moderate to severe nonrheumatic mitral stenosis.
* Currently prescribed dual antiplatelet therapy (ASA plus either clopidogrel, ticagrelor, or prasugrel) for an indication other than AF.
* Has an independent, non-AF indication for oral anticoagulation.
* Has a non-modifiable impediment to effective use of web-based tools. Examples include lack of internet access, lack of English literacy (Grade 5 level).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The 9-Item Shared Decision Making Questionnaire (SDM-Q-9: patient version). | Immediately after clinic visit
  The SDM-Q-9 is a reliable, brief and well accepted instrument for measuring shared decision-making process from the patient's perspective. The statements can be rated on a 6-point scale ranging from completely disagree (0) to completely agree (5). The addition of these scores for the 9 items will result in a score between 0 and 45. The raw score (over 45) can be converted to an equivalent number between 0 and 100 by multiplying by 20/9. 0 represents the lowest possible level of SDM while 100 corresponds to highest level of SDM.

OTHER OUTCOMES:
OPTION 5: Objective assessment of shared decision-making | Immediately after clinic visit
  The OPTION-5 tool will be used to to assess the quality of shared decision-making from an objective observer perspective. This score rates 5 key elements of SDM in the patient-clinician interaction. each on an ordinal scale from 0 (no effort) to 4 (exemplary effort), for a total possible score of 20. The score is rescaled to a range of 0 to 100, with 100 indicating exemplary effort for shared decision making. The OPTION-5 rating score will be completed by trained research personnel using audio recordings of the clinic visit.
Physician version of the 9-Item Shared Decision Making Questionnaire (SDM-Q-Doc) | Immediately after clinic visit
  The SDM-Q-9 is a reliable, brief and well accepted instrument for measuring shared decision-making process from the physician's perspective. The statements can be rated on a 6-point scale ranging from completely disagree (0) to completely agree (5). The addition of these scores for the 9 items will result in a score between 0 and 45. The raw score (over 45) can be converted to an equivalent number between 0 and 100 by multiplying by 20/9. 0 represents the lowest possible level of SDM while 100 corresponds to highest level of SDM.
Therapy decision | Immediately after clinic visit
  The patient's stated post-visit decision about stoke prevention therapy.
Decisional conflict | Immediately after clinic visit
  Using the Decisional Conflict Scale. This is a well-validated 16-item survey. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].
Visit Duration | Immediately after clinic visit
  Total visit duration, time spent discussing stroke risk, time spent reviewing decision aid results.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Wilton, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Calgary Zone, Alberta Health Services, Calgary, Alberta
  - Vita Diagnostics, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual patient data available to external researchers from this pilot study.